CLINICAL TRIAL: NCT05657457
Title: Improving Neurological Outcome for Acute Basilar Artery Occlusion With Sufficient Recanalization After Thrombectomy by Intraarterial Tenecteplase (INSIST-IT): a Prospective, Randomized, Open-label, Blinded-end Point, Multicenter Trial
Brief Title: Improving Neurological Outcome for Acute Basilar Artery Occlusion With Sufficient Recanalization After Thrombectomy by Intraarterial Tenecteplase (INSIST-IT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The interim analysis showed the potential harm of intra-arterial TNK.
Sponsor: General Hospital of Shenyang Military Region (Other)
Collaborators: Cerebrovascular Disease Collaboration & Innovation Alliance of Liaoning (Unknown)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2022) 185
Record Dates: First submitted 2022-12-02; First posted 2022-12-20 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNK group (Experimental)
  Interventions: Drug: Tenecteplase
- control group (No Intervention)

INTERVENTIONS:
Drug: Tenecteplase — intra-arterial tenecteplase
  Arms: TNK group

SUMMARY:
The potential benefit of intraarterial tenecteplase in acute basilar artery occlusion (BAO) patients with successful reperfusion following endovascular treatment (EVT) has not been studied. The current study aimed to explore the efficacy and safety of intraarterial tenecteplase in acute BAO patients with successful reperfusion after EVT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients with basilar artery occlusion who received endovascular treatment within 24 hours of estimated time of stroke onset as per BASICS trial definition;
* National Institute of Health Stroke Scale (NIHSS) ≥ 6 before endovascular treatment;
* Successful recanalization (mTICI 2b-3) after endovascular treatment;
* PC-ASPECTS ≥ 6 on CT;
* Absence of parenchymal hematoma on CT images done in the angio suite immediately after the procedure;
* Modified Rankin Scale score before stroke onset ≤ 3;
* Signed informed consent by patient or their legally authorized representative.

Exclusion Criteria:

* baseline PC ASPECTS < 5 on CT;
* More than six retrieval attempts in the same vessel;
* Hemorrhagic stroke: cerebral hemorrhage, subarachnoid hemorrhage;
* Coagulation disorders, systemic hemorrhagic diathesis, thrombocytopenia (<100000/mm3), or INR > 1.7;
* Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
* After recanalization, severe and sustained (i.e., > 5 minutes) uncontrolled hypertension (systolic blood pressure over 180mmHg or diastolic blood pressure over 105 mmHg) refractory to antihypertensive medication;
* Patients with contraindication or allergic to any ingredient of drugs in our study
* Pregnancy, plan to get pregnant or during lactation
* The estimated life expectancy is less than 6 months due to other serious diseases;
* Other conditions unsuitable for this clinical study assessed by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-05-18 (Actual); Study Completion 2025-05-18 (Actual)

PRIMARY OUTCOMES:
proportion of favorable functional outcome | Day 90
  favorable functional outcome is defined as a modified Rankin Scale (mRS) score of 0 to 3

SECONDARY OUTCOMES:
proportion of patients with an improved modified thrombolysis in cerebral infarction score | immediately after intraarterial TNK administration or at the end of endovascular treatment
the proportion of patients with modified Rankin Score (mRS) 0 to 1 | Day 90
  mRS scores range from 0 to 6: 0, no symptoms, 1 = symptoms without clinically significant disability, 2 = slight disability, 3 = moderate disability, 4 = moderately severe disability, 5 = severe disability; and 6 = death.
the proportion of patients with modified Rankin Score (mRS) 0 to 2 | Day 90
  mRS scores range from 0 to 6: 0, no symptoms, 1 = symptoms without clinically significant disability, 2 = slight disability, 3 = moderate disability, 4 = moderately severe disability, 5 = severe disability; and 6 = death.
ordinal distribution of modified Rankin Score (mRS) | Day 90
  mRS scores range from 0 to 6: 0, no symptoms, 1 = symptoms without clinically significant disability, 2 = slight disability, 3 = moderate disability, 4 = moderately severe disability, 5 = severe disability; and 6 = death.
change in modified Rankin Score (mRS) compared with premorbid mRS | Day 90
  mRS scores range from 0 to 6: 0, no symptoms, 1 = symptoms without clinically significant disability, 2 = slight disability, 3 = moderate disability, 4 = moderately severe disability, 5 = severe disability; and 6 = death.
change in National Institute of Health stroke scale (NIHSS) | 24 (-6/+24) hours
  NIHSS scores range from 0 to 42, with higher scores indicating more severe neurological deficit
proportion of early neurological improvement | 24 (-6/+24) hours
  early neurological improvement is defined as a NIHSS decrease ≥4
change in the cerebral circulation time | immediately after tenecteplase
the occurrence rate of composite events of recurrent stroke, cardiovascular or cerebrovascular events | Day 90
proportion of sympomatic intracranial hemorrhage | 24 (-6/+24) hours
  sympomatic intracranial hemorrhage is defined as a NIHSS increase ≥4 caused by intracranial hemorrhage
proportion of intraparenchymal hemorrhage | 24 (-6/+24) hours
  intraparenchymal hemorrhage was defined as confluent bleeding occupying and causing mass effect
the percentage of severe adverse events | 24 (-6/+24) hours
cerebral edema | 24 (-6/+24) hours
  cerebral edema was measure by the mount of midline shift of the brain on neuroimaging
all-cause mortality | 10 days
the number of tenecteplase infusions interrupted due to suspected active bleeding | during endovascular treatment (up to 2 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided